CLINICAL TRIAL: NCT04745806
Title: A Prospective, Single Arm, Post Marketing Study for Evaluating the Effectiveness of ActiGraft in Treating Lower Extremity Hard to Heal Wounds
Brief Title: Post Marketing Trial for Evaluating the Effectiveness of ActiGraft in Treating Lower Extremity Hard To Heal Wounds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: RedDress Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD007
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Wounds
Keywords: Chronic; Ulcer; Lower extremity; DFU; VLU
MeSH Terms: conditions — Wounds and Injuries; Bronchiolitis Obliterans Syndrome; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ActiGraft (Experimental): Whole blood clot (WBC) gel
  Interventions: Device: ActiGraft

INTERVENTIONS:
Device: ActiGraft — Whole blood clot (WBC) gel

SUMMARY:
The study is a prospective, single arm, post- marketing study. The subjects enrolled to the study will receive weekly applications of ActiGraft until complete healing or until investigator's decision that patient can no longer benefit from the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age
2. Patient with a chronic lower extremity ulcer (i.e DFU, VLU, …)
3. Ulcer duration >30 days.
4. Ulcer size decreased in less than 30% in the 14 days prior to enrollment, while treated with standard of care (or advanced treatment)
5. Subject must be willing to comply with the protocol including having blood drawn to create the ActiGraft
6. Subject can read and understand the Informed Consent form

Exclusion Criteria:

1. Presence of active underlying osteomyelitis.
2. Known malignancy in the reference wound bed or margins of the wound
3. Cannot withdraw blood in the required amount technically.
4. Subject is receiving (i.e., within the past 30 days) systemic steroids (more than 10mg per day)
5. Subject has been treated with wound dressings that include growth factors, engineered tissues or skin substitutes (within the past 30 days).
6. Subject has been treated with hyperbaric oxygen, wound VAC or Ozone gas(O3) within the past 5 days or is scheduled to receive during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Percent of Reduction in Wound Size Over 12 Weeks | 4, 8, and 12 weeks
  The change in wound area (decrease or increase) with respect to the area at baseline, expressed as a percentage.

SECONDARY OUTCOMES:
Number of Participants Achieving a Complete Wound Closure at 12 Weeks | 12 weeks
  Skin re-epithelialization without drainage or dressing requirements.
Number of Participants Achieving a Complete re-epithelialization at 18 and 24 Weeks | 18 and 24 weeks
  Skin re-epithelialization without drainage or dressing requirements.
Percent of Reduction in Wound Size Over 18 and 24 Weeks. | 18 and 24 weeks
  The change in wound area (decrease or increase) with respect to the area at baseline, expressed as a percentage for wound treated beyond 12 weeks, per the investigator's decision
The change in wound pain by 12 weeks | 12 weeks
  Pain assessment would be done by using the Numeric Rating Scale (NRS). Subject chooses a number on a 1 to 10 scale that best describes his ulcer pain, while 0 represents "No Pain" and 10- " Worst Pain Imaginable "test, a scale between .

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Sirota, Study Director — RedDress Ltd.
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Yes
The results will be part of several scientific publications.
Supporting Information: Study Protocol
Time Frame: Upon publication.